CLINICAL TRIAL: NCT01768000
Title: The Family CAT (Cognitive Adaptation Training Manual): A Test of Effectiveness
Brief Title: The Family Cognitive Adaptation Training Manual: A Test of Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Sean Kidd, Independent Clinician Scientist and Head Psychology Service, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 173/2012
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Psychosis
Keywords: Psychosis; Psychosis NOS; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Cognitive Adaptation Training (Experimental): Participants in this group will receive the Family CAT manual and DVD
  Interventions: Behavioral: Family Cognitive Adaptation Training
- Control group (No Intervention): Participants in this arm will support their family members as usual, and will not receive the Family CAT manual and DVD provided to those in the experimental arm of the study.

INTERVENTIONS:
Behavioral: Family Cognitive Adaptation Training — Family CAT is a 4 month manualised intervention designed to be administered by families independent of clinician support. A self scoring checklist is provided to assess and tailor Family CAT to the individual, along with descriptions of strategies for bathing, dressing, dental hygiene, make-up, toileting, housekeeping/care of living quarters, laundry, grocery shopping, transportation, management of money and consumables, medication management, social skills, communication and telephone use, leisure skills, work skills, and orientation. Family members will watch the DVD to gain insight into how the strategies can be implemented in real world settings. Having identified the areas of need, family members will administer the interventions and evaluate their effectiveness for the individual.
  Other Names: Family CAT
  Arms: Family Cognitive Adaptation Training

SUMMARY:
The purpose of this study is to examine the effectiveness of family cognitive adaptation training, including its impact on functioning and caregiver burden. Families that receive the manual will be compared with a control group of families that will not receive the manual. The larger goal is to add to the tools family members have access to better support their family members with schizophrenia.

DETAILED DESCRIPTION:
Efforts to address the cognitive impacts of schizophrenia can be broadly defined as falling into either compensatory or restorative categories. Restorative interventions, such as cognitive remediation, have shown promise in reducing cognitive deficits and improving functional outcomes (McGurk et al., 2007). In contrast, compensatory approaches such as Cognitive Adaptation Training work around cognitive deficits by changing the client's natural environment to support improved functioning. These compensatory strategies serve to bypass cognitive deficits and negative symptoms by organizing belongings and creating reminders and environmental cues to support specific adaptive behaviors. An example includes the individual packaging of clothes to be worn by day, to simplify the process of choosing what to wear and decrease the likelihood of clients impulsively putting on too many clothes or otherwise dressing in a manner that is not a good fit for the climate or social settings (Draper et al., 2009; Maples & Velligan, 2008).

Cognitive Adaptation Training (CAT) is a manualized intervention that was developed to help individuals compensate for the cognitive deficits associated with schizophrenia. CAT interventions commence with a neuropsychological assessment of clients to determine the best profile of strategies to be implemented for the specific cognitive classification within which the person is placed. Interventions are based on two dimensions 1) level of executive functioning (as determined by scores on a set of neurocognitive tests) and 2) whether the behaviour of the individual is characterized more by apathy (poverty of speech and movement and difficulty initiating behaviours), disinhibition (distractibility and impulsivity) or a combination of the two. Clinicians then develop and implement an individualized set of strategies that address key domains such as hygiene, safety, dress, and medication. These strategies are then altered for strengths or weaknesses in the areas of attention, memory, and fine motor skills. For example, for someone with poor attention, the colour of signs can be changed regularly or florescent colours can be used to capture attention. For someone with memory problems (particularly those with good auditory attention) audiotapes can be used to sequence behaviour.

CAT interventions are established and maintained in the home during monthly to weekly visits from a CAT therapist/trainer with the intervention typically lasting 9 months in most of the trials that have taken place to date

Outcomes of randomized trials of CAT have been promising. Compared to control conditions, clients receiving CAT have lower levels of symptomatology, lower relapse rates, higher levels of adaptive functioning, better quality of life, and better medication adherence (Velligan et al., 2000; 2002; 2007; 2008a; 2008b). In general, CAT has been shown to be beneficial for individuals with schizophrenia who vary both in degree and type of functional impairment.

The support and involvement of family in the care of individuals with schizophrenia is both one of the most important contributors to wellness and recovery and is also, unfortunately, one of the least acknowledged components of the recovery process. A high proportion of persons with severe mental illness stay in touch with family and the involvement of family in care has been associated with better clinical outcomes, improved quality of life, and less use of hospitalization (e.g., Fischer et al., 2008). Despite evidence of the importance of family in the recovery process, the contribution of family is often not adequately appreciated by treatment providers, and contact with providers is often limited. Similarly under-developed are evidence-based tools to assist families in their efforts to support the recovery of their loved ones.

It is within this context that the development of a family member version of CAT is a very promising avenue to explore. While some elements of CAT require or are otherwise optimized by administration by a mental health professional (e.g., neuropsychological testing; targeting interventions based upon ongoing clinical evaluation), there are many standard components of CAT that can be readily implemented by a family member or other key support. Examples include CAT interventions such as visual reminders regarding medication, arranging cleaning supplies in the kitchen to reinforce cleaning routines, and assisting in the use of a calendar for scheduling. We have developed a tool that facilitates family members implementing CAT components that do not require professional administration.

The initial 'beta' version of Family CAT was developed in close collaboration between Dr. Velligan's team at the University of Texas, the group implementing CAT at the CAMH site led by Dr. Kidd, and CAMH Social Workers. This 'beta' version is currently in the process of having its content reviewed by 6 families to obtain feedback regarding how readily it can be understood. Based on this feedback, we will make edits and produce the final version to be used in the trial proposed in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* the key family member/support is actively involved in the support of the individual with schizophrenia and regularly visits them (i.e., once a week or more frequently) in their home environment
* the individual being supported is identified (self-identified and identified by the family member) as having a primary diagnosis of schizophrenia
* the individual with schizophrenia is not in crisis or experiencing other forms of instability (e.g., imminent loss of housing) per verbal report that would threaten the implementation of the manual strategies
* proficiency in English

Exclusion criteria:

- none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Kidd, Ph.D, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alphs LD, Summerfelt A, Lann H, Muller RJ. The negative symptom assessment: a new instrument to assess negative symptoms of schizophrenia. Psychopharmacol Bull. 1989;25(2):159-63. No abstract available. PMID 2602512
- [Background] Byerly MJ, Nakonezny PA, Rush AJ. The Brief Adherence Rating Scale (BARS) validated against electronic monitoring in assessing the antipsychotic medication adherence of outpatients with schizophrenia and schizoaffective disorder. Schizophr Res. 2008 Mar;100(1-3):60-9. doi: 10.1016/j.schres.2007.12.470. Epub 2008 Feb 5. PMID 18255269
- [Background] Draper ML, Stutes DS, Maples NJ, Velligan DI. Cognitive adaptation training for outpatients with schizophrenia. J Clin Psychol. 2009 Aug;65(8):842-53. doi: 10.1002/jclp.20612. PMID 19521972
- [Background] Fischer EP, McSweeney JC, Pyne JM, Williams DK, Naylor AJ, Blow FC, Owen RR. Influence of family involvement and substance use on sustained utilization of services for schizophrenia. Psychiatr Serv. 2008 Aug;59(8):902-8. doi: 10.1176/ps.2008.59.8.902. PMID 18678688
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] McGurk SR, Mueser KT. Cognitive functioning, symptoms, and work in supported employment: a review and heuristic model. Schizophr Res. 2004 Oct 1;70(2-3):147-73. doi: 10.1016/j.schres.2004.01.009. PMID 15329293
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] Reichenberg A, Harvey PD. Neuropsychological impairments in schizophrenia: Integration of performance-based and brain imaging findings. Psychol Bull. 2007 Sep;133(5):833-58. doi: 10.1037/0033-2909.133.5.833. PMID 17723032
- [Background] Test MA, Greenberg JS, Long JD, Brekke JS, Burke SS. Construct validity of a measure of subjective satisfaction with life of adults with serious mental illness. Psychiatr Serv. 2005 Mar;56(3):292-300. doi: 10.1176/appi.ps.56.3.292. PMID 15746503
- [Background] van Wijngaarden B, Schene AH, Koeter M, Vazquez-Barquero JL, Knudsen HC, Lasalvia A, McCrone P. Caregiving in schizophrenia: development, internal consistency and reliability of the Involvement Evaluation Questionnaire--European Version. EPSILON Study 4. European Psychiatric Services: Inputs Linked to Outcome Domains and Needs. Br J Psychiatry Suppl. 2000;(39):s21-7. doi: 10.1192/bjp.177.39.s21. PMID 10945074
- [Background] Velligan DI, Bow-Thomas CC, Huntzinger C, Ritch J, Ledbetter N, Prihoda TJ, Miller AL. Randomized controlled trial of the use of compensatory strategies to enhance adaptive functioning in outpatients with schizophrenia. Am J Psychiatry. 2000 Aug;157(8):1317-23. doi: 10.1176/appi.ajp.157.8.1317. PMID 10910797
- [Background] Velligan DI, Prihoda TJ, Ritch JL, Maples N, Bow-Thomas CC, Dassori A. A randomized single-blind pilot study of compensatory strategies in schizophrenia outpatients. Schizophr Bull. 2002;28(2):283-92. doi: 10.1093/oxfordjournals.schbul.a006938. PMID 12693434
- [Background] Velligan DI, Lam F, Ereshefsky L, Miller AL. Psychopharmacology: Perspectives on medication adherence and atypical antipsychotic medications. Psychiatr Serv. 2003 May;54(5):665-7. doi: 10.1176/appi.ps.54.5.665. No abstract available. PMID 12719495
- [Background] Velligan DI, Diamond PM, Mintz J, Maples N, Li X, Zeber J, Ereshefsky L, Lam YW, Castillo D, Miller AL. The use of individually tailored environmental supports to improve medication adherence and outcomes in schizophrenia. Schizophr Bull. 2008 May;34(3):483-93. doi: 10.1093/schbul/sbm111. Epub 2007 Oct 10. PMID 17932089
- [Background] Velligan DI, Diamond PM, Maples NJ, Mintz J, Li X, Glahn DC, Miller AL. Comparing the efficacy of interventions that use environmental supports to improve outcomes in patients with schizophrenia. Schizophr Res. 2008 Jul;102(1-3):312-9. doi: 10.1016/j.schres.2008.02.005. Epub 2008 Apr 18. PMID 18374542
- [Derived] Kidd SA, Kerman N, Ernest D, Maples N, Arthur C, de Souza S, Kath J, Herman Y, Virdee G, Collins A, Velligan D. A pilot study of a family cognitive adaptation training guide for individuals with schizophrenia. Psychiatr Rehabil J. 2018 Jun;41(2):109-117. doi: 10.1037/prj0000204. Epub 2016 Aug 22. PMID 27547853
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca/en/research/Pages/research.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited between March 2013 and February 2014 in Ontario, Canada.
Groups:
- Family Cognitive Adaptation Training - Caregivers; Family Cognitive Adaptation Training - Family Members: Participants in this group will receive the Family CAT manual and DVD.
  Family Cognitive Adaptation Training: Family CAT is a 4 month manualised intervention designed to be administered by families independent of clinician support. A self scoring checklist is provided to assess and tailor Family CAT to the individual, along with descriptions of strategies for bathing, dressing, dental hygiene, make-up, toileting, housekeeping/care of living quarters, laundry, grocery shopping, transportation, management of money and consumables, medication management, social skills, communication and telephone use, leisure skills, work skills, and orientation. Family members will watch the DVD to gain insight into how the strategies can be implemented in real world settings. Having identified the areas of need, family members will administer the interventions and evaluate their effectiveness for the individual.
- Control Group - Caregivers; Control Group - Family Members: Participants in this arm will support their family members as usual, and will not receive the Family CAT manual and DVD provided to those in the experimental arm of the study.
Period: Overall Study
Arm/Group | Family Cognitive Adaptation Training - Caregivers | Control Group - Caregivers | Family Cognitive Adaptation Training - Family Members | Control Group - Family Members
Started | 10 | 10 | 10 | 10
Completed | 9 | 8 | 9 | 8
Not Completed | 1 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Analysis includes all participants recruited into the study that completed the entire baseline assessment.
Groups:
- Family Cognitive Adaptation Training - Family Members; Family Cognitive Adaptation Training - Caregivers: Participants in this group will receive the Family CAT manual and DVD.
  Family Cognitive Adaptation Training: Family CAT is a 4 month manualized intervention designed to be administered by families independent of clinician support. A self scoring checklist is provided to assess and tailor Family CAT to the individual, along with descriptions of strategies for bathing, dressing, dental hygiene, make-up, toileting, housekeeping/care of living quarters, laundry, grocery shopping, transportation, management of money and consumables, medication management, social skills, communication and telephone use, leisure skills, work skills, and orientation. Family members will watch the DVD to gain insight into how the strategies can be implemented in real world settings. Having identified the areas of need, family members will administer the interventions and evaluate their effectiveness for the individual.
- Total: Total of all reporting groups
Arm/Group | Family Cognitive Adaptation Training - Family Members | Family Cognitive Adaptation Training - Caregivers | Control Group - Family Members | Control Group - Caregivers | Total
Number analyzed (Participants) | 10 | 10 | 9 | 9 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 9 | 8 | 36
  >=65 years | 0 | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 4 | 6 | 19
  Male | 8 | 3 | 5 | 3 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Asian East | 1 | 1 | 0 | 0 | 2
  Asian South | 1 | 3 | 1 | 0 | 5
  Asian South East | 1 | 0 | 0 | 0 | 1
  Black Canadian | 1 | 0 | 1 | 1 | 3
  Latin American | 0 | 1 | 0 | 0 | 1
  White Canadian | 5 | 5 | 5 | 3 | 18
  White European | 0 | 0 | 1 | 3 | 4
  Other | 0 | 0 | 0 | 1 | 1
  Asian (not specified) | 0 | 0 | 1 | 1 | 2
  Not specified | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 9 | 9 | 38
Employment status [Number; unit: participants]
  Full-time | 1 | 4 | 1 | 4 | 10
  Part-time | 1 | 2 | 1 | 3 | 7
  In school | 3 | 0 | 1 | 0 | 4
  Unemployed | 5 | 1 | 5 | 1 | 12
  Retired | 0 | 0 | 1 | 0 | 1
  Contract work | 0 | 3 | 0 | 0 | 3
  Not specified | 0 | 0 | 0 | 1 | 1
Level of education [Number; unit: participants]
  Completion of graduate school | 0 | 2 | 0 | 2 | 4
  Completion of undergraduate university/college | 0 | 5 | 2 | 4 | 11
  Partial undergraduate university/college | 7 | 2 | 5 | 0 | 14
  Completion of high school | 1 | 1 | 1 | 2 | 5
  Partial high school | 1 | 0 | 1 | 0 | 2
  Not specified | 1 | 0 | 0 | 1 | 2
Housing [Number; unit: Participants] — Housing data was collected only for the participant with psychosis and NOT the family member.
  Participants
    Own/rent apartment or home | 0 | NA — Housing data was collected only for the participant with psychosis and NOT the family member. | 2 | NA — Housing data was collected only for the participant with psychosis and NOT the family member. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Supported housing | 1 | NA — Housing data was collected only for the participant with psychosis and NOT the family member. | 1 | NA — Housing data was collected only for the participant with psychosis and NOT the family member. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Live with family | 9 | NA — Housing data was collected only for the participant with psychosis and NOT the family member. | 6 | NA — Housing data was collected only for the participant with psychosis and NOT the family member. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Multnomah Community Ability Scale (MCAS)
Description: The Multnomah Community Ability Scale (MCAS; Barker et al., 1994) is a 17-item scale assessing functionality in four domains - health, adaptation, social skills and behaviour. Ratings are made on the basis of an interview with the patient and their family member. The MCAS generates a total score ranging from 17 to 85. Items on the MCAS are scored on a five-point scale. The four total domain scores ranges are - health, 5-25; adaptation, 3-15; social skills, 5-25; behaviour, 4-20. Lower ratings indicate less ability. Higher ratings usually mean an assessment of greater ability.
Time Frame: 4 months following baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family Cognitive Adaptation Training - Caregivers | Control Group - Caregivers | Family Cognitive Adaptation Training - Family Members | Control Group - Family Members
Number analyzed (Participants) | 9 | 9 | 8 | 8
units on a scale
  Total | 67.78 (5.70) | 74.63 (5.45) | 70.00 (5.10) | 74.38 (5.15)
  Health | 21.67 (2.34) | 22.13 (2.36) | 21.56 (1.88) | 21.50 (1.93)
  Adaptation | 10.89 (2.57) | 13.25 (1.67) | 11.78 (1.92) | 13.00 (1.69)
  Social Skills | 17.44 (3.17) | 20.63 (2.50) | 18.33 (3.87) | 20.75 (2.71)
  Behaviour | 17.78 (1.72) | 18.63 (1.77) | 18.33 (1.80) | 19.13 (1.36)

2. Secondary Outcome: Brief Adherence Rating Scale (BARS)
Description: The Brief Adherence Rating Scale (BARS; Byerly et al., 2008) is a 4-item, valid, reliable, sensitive, measure with which to obtain specific estimates of antipsychotic medication adherence of outpatients with schizophrenia. A total percentage score on a scale ranging from 0 to 100, with 0 indicating less adherence and 100 total adherence.
Time Frame: 4 months following baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family Cognitive Adaptation Training - Caregivers | Control Group - Caregivers | Family Cognitive Adaptation Training - Family Members | Control Group - Family Members
Number analyzed (Participants) | 9 | 9 | 8 | 8
units on a scale | 77.22 (35.98) | 87.50 (35.36) | 59.33 (44.03) | 88.75 (31.82)

3. Secondary Outcome: Satisfaction With Life Scale
Description: 8 out of 18 items from the Satisfaction With Life Scale (Test et al., 2005) will measure the perceived quality of life of the individual with schizophrenia by tapping into global satisfaction in domains relevant to CAT (e.g., How satisfied are you with yourself on the whole? - 5 point scale, not at all - great deal). This scale is well-validated with a schizophrenia population and is being shortened as not all items are relevant to CAT nor expected to be sensitive to change in a 4 month period, and there is a need to abbreviate the battery to reduce the risk of fatigue in a lengthy phone interview. These 8 items comprise four domains of social relationships, employment/work, social and present life and living situation. A low score indicates less satisfaction in these domains and a higher score indicating greater satisfaction. Total scores can range from 8-40 and subscale scores range from 1-5.
Time Frame: 4 months following baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family Cognitive Adaptation Training - Family Members | Control Group - Family Members
Number analyzed (Participants) | 9 | 8
units on a scale
  Social Relationships | 2.06 (0.92) | 2.18 (0.73)
  Employment/Work | 1.63 (1.16) | 2.17 (0.41)
  Social & Present Life | 2.00 (0.99) | 2.29 (0.76)
  Living Situation | 3.11 (0.49) | 3.00 (0.66)

4. Secondary Outcome: Involvement Evaluation Questionnaire (IES)
Description: The 31-item Involvement Evaluation Questionnaire (IEQ; Van Wijngaarden et al., 2000) measures caregiver burden. It has been validated for caregivers of individuals with schizophrenia, covers a broad domain of caregiving consequences and refers to burden experienced within the past 4 weeks. Mean scores are calculated for the total scale and sub-scales. Total scores can range from 29 to 145 with sub-scale domains ranging - tension, 9-45; supervision, 6-30; worrying, 6-30; and urging, 8-40. Lower total and subscale scores indicate less burden and higher scores greater level of caregiver burden.
Time Frame: 4 months following baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family Cognitive Adaptation Training - Caregivers | Control Group - Caregivers
Number analyzed (Participants) | 9 | 8
units on a scale
  Total | 57.72 (9.66) | 49.25 (11.15)
  Tension | 15.50 (4.27) | 14.13 (2.85)
  Supervision | 8.22 (2.05) | 7.50 (1.07)
  Worrying | 17.89 (4.31) | 15.25 (4.40)
  Urging | 20.56 (7.13) | 16.38 (5.66)

ADVERSE EVENTS:
Arm/Group | Family Cognitive Adaptation Training - Caregivers | Control Group - Caregivers | Family Cognitive Adaptation Training - Family Members | Control Group - Family Members
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No